CLINICAL TRIAL: NCT02892123
Title: Phase I Trial of ZW25 in Patients With Locally Advanced (Unresectable) and/or Metastatic HER2-expressing Cancers
Brief Title: Trial of ZW25 (Zanidatamab) in Patients With Advanced HER2-expressing Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW25-101
Expanded Access: NCT04578444 (No longer available)
Record Dates: First submitted 2016-08-23; First posted 2016-09-08 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: HER2-expressing Cancers
Keywords: HER2; Bispecific antibody; Biparatopic antibody; Immunotherapy; Breast cancer; Gastroesophageal adenocarcinoma (GEA); Gastric cancer; Gastroesophageal junction (GEJ) cancer; Ovarian cancer; Non-small cell lung cancer (NSCLC); Chemotherapy; Paclitaxel; Capecitabine; Vinorelbine; Tucatinib
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — zanidatamab; Paclitaxel; Capecitabine; Vinorelbine; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZW25 (Zanidatamab) Monotherapy and ZW25 Combination Therapy (Experimental)
  Interventions: Drug: ZW25 (Zanidatamab); Drug: Paclitaxel; Drug: Capecitabine; Drug: Vinorelbine; Drug: Tucatinib

INTERVENTIONS:
Drug: ZW25 (Zanidatamab) — ZW25 administered IV once weekly, once every 2 weeks, or once every 3 weeks. Part 1: in multiple increasing doses; Part 2: ZW25 given at the MTD, OBD, or an RD identified in Part 1; Part 3: ZW25 given at the MTD, OBD, or an RD combined with one of the following selected drug combination:
Drug: Paclitaxel — Combination therapy with ZW25 - Part 3 Treatment Groups 1 and 4
Drug: Capecitabine — Combination therapy with ZW25 - Part 3 Treatment Groups 2 and 5
Drug: Vinorelbine — Combination therapy with ZW25 - Part 3 Treatment Groups 3 and 6
Drug: Tucatinib — Combination therapy with ZW25 and Capecitabine - Part 3 Treatment Group 7
Drug: Tucatinib — Combination therapy with ZW25 - Part 3 Treatment Group 8 (may be opened if recommended by the Safety Monitoring Committee and/or the sponsor)

SUMMARY:
This is a first-in-human, 3-part study to investigate the safety, tolerability, and effectiveness of ZW25 (zanidatamab) by itself and combined with selected chemotherapy agents in patients with locally advanced (unresectable) and/or metastatic human epidermal growth factor receptor 2 (HER2)-expressing cancers. This study will also the evaluate the way the body absorbs, distributes, and eliminates ZW25 (pharmacokinetics or PK).

DETAILED DESCRIPTION:
Part 1 of the study will evaluate increasing doses of ZW25 to find the highest dose of ZW25 that does not cause unacceptable side effects (maximum-tolerated dose or MTD), the lowest safe dose with the highest rate of effectiveness (optimal biological dose or OBD), and/or other recommended dosages (RDs) of ZW25 in up to 7 dose-specific cohorts. Eligible patients include those with selected HER2-expressing locally advanced (unresectable) and/or metastatic cancers that have progressed after receipt of all therapies known to confer clinical benefit (or ineligible to receive therapy).

Part 2 of the study will further evaluate the safety, tolerability, and efficacy of ZW25 in patients with selected HER2-expressing locally advanced (unresectable) and/or metastatic cancers that have progressed after receipt of all therapies known to confer clinical benefit (or ineligible to receive therapy) in up to 5 separate disease-specific cohorts.

Part 3 of the study will evaluate the safety, tolerability, and efficacy of ZW25 combined with selected chemotherapy agents, including paclitaxel, capecitabine, vinorelbine, or capecitabine and tucatinib. Patients with selected HER2-expressing locally advanced (unresectable) and/or metastatic cancers that have progressed after at least 1 and no more than 3 prior systemic chemotherapy regimens will be evaluated in this part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. HER2-expressing cancer as follows:

   Part 1:
   * Cohorts 1 - 3: Any locally advanced (unresectable) and/or metastatic HER2-expressing (HER2 1+, 2+, or 3+ by IHC) cancer (including but not limited to breast, gastric, ovarian, colorectal and non-small cell lung) that has progressed after receipt of all therapies known to confer clinical benefit
   * Cohort 4:

     * HER2 IHC 2+ /FISH- breast cancer or gastroesophageal adenocarcinoma (GEA)
     * HER2 IHC 3+ or HER2 IHC 2+ /FISH+ breast cancer or GEA
     * Any other HER2 IHC 3+ or FISH+ cancer

       * HER2-overexpressing (3+ by IHC) or HER2-2+ and FISH+ breast cancer must have progressed after prior treatment with trastuzumab, pertuzumab, and T-DM1
       * HER2-overexpressing (3+ by IHC) or HER2-2+ and FISH+ GEA must have progressed after prior treatment with trastuzumab
       * Patients with colorectal cancer must be KRAS wild-type
       * Patients with NSCLC must have ALK wild-type, EGFR wild-type, and ROS1 fusion negative as determined by standard methods
   * Cohorts 5 - 6: HER2 IHC 3+ or HER2 IHC 2+ /FISH+ GEA must have progressed after prior treatment with trastuzumab
   * Cohort 7 (only at selected sites): HER2 IHC 3+, HER2 IHC 2+ /FISH+, or HER2 IHC 2+ /FISH- breast cancer must have progressed after prior treatment with trastuzumab, pertuzumab, and T-DM1

   Part 2:

   Locally advanced (unresectable) and/or metastatic cancer that has progressed after receipt of all therapies known to confer clinical benefit (unless ineligible to receive a specific therapy) as follows:
   * Cohort 1: HER2 IHC 2+/FISH- breast cancer
   * Cohort 2: HER2 IHC 3+ or HER2 IHC 2+/FISH+ breast cancer
   * Cohort 3: HER2 IHC 2+/FISH- GEA
   * Cohort 4: HER2 IHC 3+ or HER2 IHC 2+/FISH+ GEA
   * Cohort 5: Any other HER2 IHC 3+ or IHC 2+/FISH+ cancer, including the following:

     * Cohort 5a: HER2 IHC 3+ or IHC 2+/FISH+ GI cancers other than GEA (patients with colorectal cancer must be KRAS wild-type.)
     * Cohort 5b: Any other HER2 IHC 3+ or IHC 2+/FISH+ solid tumor types that are not breast or GI cancers (patients with NSCLC must have ALK wild-type, EGFR wild-type, and ROS1 fusion negative as determined by standard methods; patients with ovarian cancers must be KRAS wild type.)

   Part 3:

   Locally advanced (unresectable) and/or metastatic cancer as follows:
   * HER2 IHC 1+ or IHC2+/FISH- breast cancer patients (TGs 1, 2, or 3) who have received at least 1 and no more than 3 prior systemic chemotherapy regimens
   * HER2 IHC 3+ or IHC 2+/FISH+ breast cancer patients (TGs 1, 2, or 3) who have received prior therapy with trastuzumab, pertuzumab, and T-DM1, at least 1 and no more than 3 prior systemic chemotherapy regimens
   * HER2 IHC 2+ or 3+ FISH+ or FISH- GEA patients (TGs 1 or 2) who have received at least 1 and no more than 3 prior systemic chemotherapy regimens
   * HER2 IHC 3+ or IHC 2+/FISH+ GEA patients who have received prior therapy with trastuzumab (TG4; ZW25 + paclitaxel)
   * HER2 IHC 3+, IHC 2+/FISH+ or otherwise HER2-positive per ASCO/CAP guidelines breast cancer patients who have received prior therapy with trastuzumab, pertuzumab, and T-DM1 (TG5; ZW25 + capecitabine)
   * HER2 IHC 3+, IHC 2+/FISH+ or otherwise HER2-positive per ASCO/CAP guidelines breast cancer patients (TG6) who have received prior therapy with trastuzumab, pertuzumab, and T-DM1
   * HER2 IHC 3+, IHC2+/FISH+, or otherwise HER2-positive per ASCO/CAP guidelines breast cancer patients (TG7) who have received prior therapy with trastuzumab, pertuzumab, and T-DM1
   * HER2 IHC 3+, IHC 2+/FISH+, or otherwise HER2-positive per ASCO/CAP guidelines breast cancer patients (TG8) who have received prior therapy with trastuzumab, pertuzumab, and T-DM1
2. ≥ 18 years of age
3. ECOG performance status of 0 or 1
4. Life expectancy of at least 3 months per the investigator's assessment.
5. Adequate organ function
6. Adequate cardiac left ventricular function, as defined by a LVEF >/= institutional standard of normal
7. For Part 1 Cohorts 1 - 3: evaluable disease (target or non-target lesions) per RECIST version 1.1. For Part 1 Cohorts 4 - 7, and Parts 2 and 3: measurable disease (target lesions) per RECIST version 1.1
8. Able to provide tumor sample (fresh or archived)
9. For Part 3 TGs 7 and 8 only - based on screening brain MRI, patients must have one of the following:

   * No evidence of brain metastases
   * Untreated brain metastases not needing immediate local therapy. For patients with untreated CNS lesions > 2.0 cm on screening contrast brain MRI, discussion with and approval from the medical monitor is required prior to enrollment
   * Previously treated brain metastases that are either stable since treatment or have progressed since prior local CNS therapy, provided there is no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator

Exclusion Criteria:

1. Experimental therapies within 4 weeks before first ZW25 dosing
2. Treatment with other cancer therapy not otherwise specified within 4 weeks before ZW25 dosing
3. Anthracyclines within 90 days before first ZW25 dosing or lifetime load exceeding 300 mg/m² adriamycin or equivalent
4. Trastuzumab, pertuzumab, lapatinib, or T-DM1 within 3 weeks before first ZW25 dosing
5. Patients in Part 3 TG4 must not have received prior taxanes
6. Patients in Part 3 TG5 must not have received prior capecitabine for metastatic disease or received any prior fam-trastuzumab deruxtecan-nxki (DS-8201a)
7. With the exception of Part 3 TGs 7 and 8, untreated brain metastases (patients with treated brain mets who are off steroids and are stable for at least 1 month at the time of screening are eligible)
8. Pregnant or breast-feeding women
9. History of life-threatening hypersensitivity to monoclonal antibodies or to recombinant proteins or excipients in drug formulation
10. Acute or chronic uncontrolled renal disease, pancreatitis or liver disease (with exception of patients with Gilbert's Syndrome, asymptomatic gall stones, liver metastases, or stable chronic liver disease per investigator assessment)
11. Peripheral neuropathy > Grade 2
12. Clinically significant interstitial lung disease
13. Known active hepatitis B or C or known infection with HIV
14. Immunosuppressive corticosteroids equivalent to > 15mg/day of prednisone within 2 weeks before first ZW25 dose
15. QTc Fridericia (QTcF) > 450 ms
16. Having clinically significant cardiac disease such as ventricular arrhythmia requiring therapy, uncontrolled hypertension or any history of symptomatic CHF
17. Having known myocardial infarction or unstable angina within 6 months before first ZW25 dosing
18. Patients in Part 3 TG7 must not have received prior capecitabine or tucatinib for metastatic disease
19. Patients in Part 3 TG8 must not have received prior tucatinib therapy for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who experience dose-limiting toxicities (DLTs) (Part 1) | Up to 8 months
The proportion patients who experience laboratory abnormalities and/or adverse events as defined by CTCAE v4.03 that are related to treatment (Parts 2 and 3) | Throughout the duration of the study; up to 2 years

SECONDARY OUTCOMES:
Serum concentrations of ZW25 | Throughout the duration of the study; up to 2 years
The proportion of patients who develop detectable anti-drug antibodies | Throughout the duration of the study; up to 2 years
The proportion of patients with an objective response (partial response or complete response) as defined by RECIST 1.1 criteria | Throughout the duration of the study; up to 2 years
Progression free survival as defined by RECIST 1.1 criteria | Throughout the duration of the study; up to 2 years
The proportion patients who experience laboratory abnormalities and/or adverse events as defined by CTCAE v4.03 that are related to treatment (Part 1) | Throughout the duration of the study; up to 2 years

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - USC/Norris Cancer Center, Los Angeles, California
  - Hoag Family Cancer Institute, Newport Beach, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Sarah Cannon - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Canada (3):
  - University of Ottawa, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meric-Bernstam F, Beeram M, Hamilton E, Oh DY, Hanna DL, Kang YK, Elimova E, Chaves J, Goodwin R, Lee J, Nabell L, Rha SY, Mayordomo J, El-Khoueiry A, Pant S, Raghav K, Kim JW, Patnaik A, Gray T, Davies R, Ozog MA, Woolery J, Lee KW. Zanidatamab, a novel bispecific antibody, for the treatment of locally advanced or metastatic HER2-expressing or HER2-amplified cancers: a phase 1, dose-escalation and expansion study. Lancet Oncol. 2022 Dec;23(12):1558-1570. doi: 10.1016/S1470-2045(22)00621-0. Epub 2022 Nov 16. PMID 36400106